CLINICAL TRIAL: NCT01573403
Title: Effect of DLBS2411 on Gastric pH Regulation in Healthy Volunteers : Comparison With Placebo
Brief Title: Efficacy and Safety of DLBS2411 in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLBS2411-0111
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Gastric pH Regulation in Healthy Volunteers
Keywords: Proton pump inhibitor (PPI); DLBS2411; gastric pH

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment 1 (Experimental): one dose of DLBS2411 @250 mg
  Interventions: Drug: DLBS2411
- Treatment II (Experimental): two doses of DLBS2411 @250 mg
  Interventions: Drug: DLBS2411
- Treatment III (Placebo Comparator)
  Interventions: Drug: Placebo DLBS2411

INTERVENTIONS:
Drug: DLBS2411 — 1 caplet of DLBS2411 @250 mg and 1 placebo caplet, once daily
  Arms: Treatment 1
Drug: DLBS2411 — 2 caplets of DLBS2411 @250 mg, once daily
  Arms: Treatment II
Drug: Placebo DLBS2411 — 2 placebo caplets of DLBS2411, once daily
  Arms: Treatment III

SUMMARY:
This is a 3-arm, double-blind, randomized, controlled, parallel and dose ranging clinical study for 3 days of therapy to investigate the effect of DLBS2411 in gastric pH regulation as well as its safety in healthy volunteers.

DLBS2411 has similar mechanism of action with proton-pump inhibitors (PPIs). However, it is hypothetically more potential than PPIs in suppressing gastric acid as our previous preclinical studies with DLBS2411 have proven its effects not only on the activity of H+/K+ ATPase, the enzyme that regulates proton pump in stomach, but also on its gene expression. It is hypothesized that DLBS2411 may benefit on gastric pH regulation in healthy volunteers.

DETAILED DESCRIPTION:
There will be 3 groups of treatment; each group will consist of 18 subjects with the treatment regimens :

* Treatment I : 1 caplet of DLBS2411 250 mg and 1 placebo caplet of DLBS2411, once daily
* Treatment II : 2 caplets of DLBS2411 250 mg, once daily
* Treatment III : 2 placebo caplets of DLBS2411, once daily

Clinical examination to evaluate the investigational drug's efficacy will be performed by a 24-hour-gastric pH monitoring after the first dose of study drug administration. Besides, the pH of the gastric fluid will also be measured at the end of study (Day 3 of treatment). Safety examination will be performed at baseline and at end of study. The occurrence of adverse event will be observed during the study.

All subjects will be under direct supervision of a medical doctor during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with age of 18-45 years
* Healthy as confirmed by vital signs, clinical and laboratory assessments (normal blood pressure, normal plasma glucose level, normal values of all hematological parameters, adequate liver and renal function)
* BMI 18-25 kg/m2
* Able to take oral medication

Exclusion Criteria:

* Gastric pH ≥ 4 at screening
* Currently being an active smoker and suffering from chronic alcoholism
* History of or currently peptic ulcer
* Having clinical diagnosis of Zollinger Ellison syndrome
* Taking any H2RAs, PPIs, antacids, or gastric mucosal protectors within 2 weeks prior to screening
* Taking any other medicines, supplements, or herbals within 3 days prior to screening
* History of gastro-intestinal disturbances necessitating long-term treatment with any acid suppressing medication, antacids, or gastric mucosal protectors
* The presence of any chronic diseases
* Currently being afflicted by serious infection(s)
* Participation in any other clinical studies within 30 days prior to screening

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Percentage of time over 24 hours during which gastric pH is > 4 | 24 hours
  Percentage of time over 24 hours during which gastric pH is > 4 after a single dose of study medication

SECONDARY OUTCOMES:
The onset of action | 24 hours
  The onset of action, which is defined as time taken to achieve gastric pH of > 4 after the initial dose of study medication
24-hour median gastric pH | 24 hours
  24-hour median gastric pH after the initial dose of study medication
Gastric pH at the end of study | 3 days
  Gastric pH after a repeated (3-day) dosing of study medication
Change of ECG description from baseline | baseline and 3 days after treatment initiation
  ECG will be evaluated at baseline (Day 1st)and at end of study (Day 3rd)
Routine haematology | Baseline and 3 days after treatment initiation
  Routine haematology (hemoglobin level, hematocrit, erythrocyte count, leucocyte count, differentiation of WBC and platelet count) will be evaluated at baseline and at end of study (Day 3rd)
Liver function | baseline and 3 days after treatment initiation
  Liver function (ALT, AST, γ-GT, and total bilirubin levels) will be evaluated at baseline and at end of study (Day 3rd)
Renal function | Baseline and 3 days after treatment initiation
  Renal function (serum creatinine level) will be evaluated at baseline and at end of study (Day 3rd)
Urinalysis parameters | Baseline and 3 days after treatment initiation
  Urinalysis parameters (urine color, pH, presence of glucose, protein, sediments, epithelial cells, erythrocyte, leucocyte, and others) will be evaluated at baseline and at end of study (Day 3rd)
Adverse events | 3 days or until all adverse events have been recovered or stabilized (which ever comes first)
  Type and number of adverse events as well as number of subjects experiencing the events will be observed and evaluated during study period (3 days of treatment)and until the end of study or all adverse events have been recovered or stabilized (which ever comes first).

CONTACTS AND LOCATIONS:
Overall Officials: Murdani Abdullah, Dr., dr., SpPD-KGEH, Principal Investigator — Division of Gastroenterology, Department of Internal Medicine, Faculty of Medicine, University of Indonesia, dr. Cipto Mangunkusumo Hospital, Jakarta Indonesia
Locations (1):
- Division of Gastroenterology, Department of Internal Medicine, dr. Cipto Mangunkusumo Hospital, Jakarta Center, Jakarta Special Capital Region, Indonesia